CLINICAL TRIAL: NCT04477798
Title: Protein Classifier for Thyroid Indeterminate Nodules： a Multi-center Prospective Clinical Study
Brief Title: Protein Classifier for Thyroid Indeterminate Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luo Dingcun (Other)
Responsible Party: Sponsor-Investigator, Luo Dingcun, vice president of hospital, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZhejiangU20200701
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCT-DIA/MS (Experimental): PCT-DIA/MS protein classifier supported by artificial neural networks will be validated to classify thyroid indeterminate nodules
  Interventions: Diagnostic Test: PCT-DIA/MS

INTERVENTIONS:
Diagnostic Test: PCT-DIA/MS — PCT-DIA/MS will be validated to classify FNA biopsy specimens

SUMMARY:
In multi-center, prospective, double-blind cohorts, PCT-DIA/MS protein classifier supported by artificial neural networks will be validated to classify thyroid indeterminate nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with aged 18 to 70 years old;
2. Patients with thyroid nodules who have not been treated with drugs;
3. Patients who were diagnosed as Bethesda III and IV by cytology and pathology before operation;
4. Patients who underwent total / partial thyroidectomy and had histopathological reports of corresponding cellular pathological punctured nodules;
5. Patients voluntarily participate in the study after informed consent.

Exclusion Criteria:

1. Patients without operation;
2. Patients with insufficient FNA sample size (judged by the laboratory).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
protein classifier | immediately after the procedure
  classify thyroid indeterminate nodules as Benign or Malignant

CONTACTS AND LOCATIONS:
Overall Officials: Dingcun Luo, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital Affiliated to Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No